CLINICAL TRIAL: NCT06700096
Title: An Open-Label, Comparative Study of the Efficacy, Safety and Pharmacodynamics of Single Dose of ANB-002 in Patients With Hemophilia B
Acronym: MAGNOLIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANB-002-2
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lead-in (No Intervention): All subjects will be enrolled in the Lead-in period in order to collect information on individual bleeding rate anf FIX concentrates consumption
- ANB-002 (arvenacogene sanparvovec) (Experimental): After completion of lead-in period subjects will enter the main period which starts with ANB-002 (arvenacogene sanparvovec) infusion.
  Interventions: Genetic: ANB-002

INTERVENTIONS:
Genetic: ANB-002 — Adeno-associated viral vector carrying the FIX gene single infusion
  Other Names: arvenacogene sanparvovec
  Arms: ANB-002 (arvenacogene sanparvovec)

SUMMARY:
The aim of the study is to demonstrate non-inferiority of ANB-002 compared with preventive use of coagulation factor IX (FIX) in adult subjects with hemophilia B with FIX activity ≤2% and without FIX inhibitor. The study will have an open-label single-arm design.

DETAILED DESCRIPTION:
After signing the ICF and screening examination the subjects are to be included in the Non-interventional lead-in period in which the subject will receive standard FIX prevention. The lead-in period will last for at least 6 month for every subject.

After completiong the lead-in period subjects will enter the main (interventional) period.

At the first visit of the main period subjects will recieve investigational product ANB-002.

The main period ends 18 months after the administration of ANB-002, after which subjects will switch to the follow-up period and will be evaluated up to 5 years after the ANB-002 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with hemophilia B aged 18 or older
* FIX activity ≤2%
* Absense of FIX inhibitor
* ≥150 previous exposure days of treatment with FIX concentrates

Exclusion Criteria:

* Any diseases of blood and hematopoietic organs other than hemophilia B
* A history of any gene therapy, including ANB-002
* Diagnosed HIV-infection, not controlled with anti-viral therapy
* Active HBV or HCV infection
* Anti-AAV5 antibodies
* Any active systemic infections or recurrent infections requiring systemic therapy
* Any other disorders associated with severe immunodeficiency
* Relevant hepatic disorders or conditions that can be a symptom of existing liver disorder
* Malignancies with less than 5 years of remission

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate (ABR) before and after a single dose of ANB-002 | Lead-in period: at least 6 months prior to ANB-002 infusion (Lead-in arm); Month 12 to Month 18 post infusion (ANB-002 arm)
  A comparison will be made between the mean ABR values in the lead-in period and within 12 months after stabilization of endogenous FIX activity, but not later than 18 months after the ANB-002 dose

SECONDARY OUTCOMES:
FIX activity | 18 months after drug administration; final assessment - 5 years
Annualized FIX consumption | 18 months after drug administration; final assessment - 5 years
Proportion of subjects not receiving FIX prevention | 18 months after drug administration
Annualized bleeding rate (ABR) | 18 months after drug administration; final assessment - 5 years
Proportion of subjects with spontaneous bleedings | 18 months after drug administration; final assessment - 5 years
Annualized rate of spontaneous bleedings | 18 months after drug administration; final assessment - 5 years
Proportion of subjects with hemarthrosis | 18 months after drug administration; final assessment - 5 years
Annualized hemarthrosis rate | 18 months after drug administration; final assessment - 5 years
Proportion of subjects with bleedings requiring FIX concentrate therapy | 18 months after drug administration; final assessment - 5 years
Annualized rate of bleedings requiring therapy with FIX concentrates | 18 months after drug administration; final assessment - 5 years
Proportion of subjects without bleeding within 12 months after stabilization of endogenous FIX activity | 12 months after stabilization of endogenous FIX activity
Proportion of subjects achieving clinical response | 18 months after drug administration
  Clinical Response is defined as FIX activity 5-150%
Proportion of subjects achieving a normalized response | 18 months after drug administration
  Normalized response is defined as FIX activity 50-150%

OTHER OUTCOMES:
Proportion of subjects with adverse reactions | 18 months after drug administration; final assessment - 5 years
Haemo-A-QoL (Hemophilia-Specific Quality of Life) score | 18 months after drug administration; final assessment - 5 years
  Haemo-A-QoL is a quality of life (QoL) assessment instrument for patients with haemophilia, including the domains of consequences of bleeding, emotional impact, physical functioning, role functioning, treatment concern, and worry. Using scale overall score ranges from 0 to 100.The high score represent low quality of life.
EuroQol-5D-3L (European Quality of Life Questionnaire) score | 18 months after drug administration; final assessment - 5 years
  The EQ-5D-5L descriptive system of health-related QoL states consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The EQ-5D-5L VAS overall score ranges from 0 to 100. A higher score is considered to be more favorable.
SF-36 (Short Form-36) score | 18 months after drug administration; final assessment - 5 years
  SF-36 is a questionnaire for evaluating health-related QoL (Quality of Life). The 36 questions are meant to reflect 8 domains of health, including physical functioning, physical role, pain, general health, vitality, social function, emotional role, and mental health. SF-3 overall score ranges from 0 to 100. The lower the score the more disability
Evaluation of the condition of joints based on the Hemophilia Joint Health Score (HJHS) | 18 months after drug administration; final assessment - 5 years
  Hemophilia Joint Health Score (HJHS) is the assessment system of joints in patients with haemophilia. Each joint (knee, elbow and ankle) receives a numeric score, which can be compared to itself over time to determine whether a joint is showing degeneration. The maximum score for an individual index joint is 20. Gait is scored 0 to 4. The maximum HJHS total score is 124, with a higher score indicating worse joint health.

CONTACTS AND LOCATIONS:
Overall Officials: Arina Arina V Zinkina-Orikhan, Study Director — Biocad
Locations (14):
- Russia (11):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Federal State Budgetary Organization of Science "Kirov Research Institute of Hematology and Blood Transfusions of Federal Medical Biological agency", Kirov
  - Federal State Budgetary Institution "National Medical Research Centre for Hematology" of the Ministry of Health of Russian Federation (Department of Clinical Diagnostics for Hematology and Hemostasis Disorders), Moscow
  - Federal State Budgetary Institution "National Medical Research Centre for Hematology" of the Ministry of Health of Russian Federation (Department of Traumatology and Reconstructive and Restorative Orthopedics for Patients with Hemophilia), Moscow
  - Federal Budgetary Institution "Moscow City Clinical Hospital named after S. P. Botkin", Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - State budgetary healthcare institution Leningrad Regional Clinical Hospital, Saint Petersburg
  - Russian Research Institute of Hematology and Transfusiology Federal State Institution of Federal Medical and Biological Agency, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Healthcare of the Russian Federation, Samara
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Healthcare of the Russian Federation, Ufa
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No